CLINICAL TRIAL: NCT00872365
Title: Effect of Micronutrients and Exercise During Pregnancy on Factors Related With Non-Transmissible Chronic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Valle, Colombia (Other)
Collaborators: Fundación FES (Other); Fundación Cardiovascular de Colombia (Other); Instituto Nacional de Salud (Unknown); University College, London (Other)
Responsible Party: Principal Investigator, Robinsón Ramírez, principal investigator, Universidad del Valle, Colombia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: Colciencias 110645921540
Record Dates: First submitted 2009-03-27; First posted 2009-03-31 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Preeclampsia; Pregnancy; Micronutrients; Exercise
Keywords: Pregnancy; Exercise; Nutrition; Micronutrients; non-transmissible chronic diseases; Endothelium
MeSH Terms: conditions — Pre-Eclampsia; Motor Activity | interventions — Micronutrients; Methods; Activities of Daily Living

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Other): Regular aerobic physical exercise + placebo
  Interventions: Behavioral: Regular aerobic physical exercise
- 2 (Other): Activities of daily living + Micronutrients
  Interventions: Dietary Supplement: Micronutrients
- 3 (Other): Regular aerobic exercise + micronutrients
  Interventions: Behavioral: Regular aerobic physical exercise; Dietary Supplement: Micronutrients
- 4 (Placebo Comparator): Activities of daily living + placebo
  Interventions: Other: Activities of daily living + placebo

INTERVENTIONS:
Behavioral: Regular aerobic physical exercise — Walking (10 minutes), aerobic exercise (30 minutes), stretching (10 minutes) and relaxation exercise (10 minutes). Exercise will be performed at three sessions per week. All sessions will be supervised by a physical therapist and a physical educator.
  Other Names: Intervention I
  Arms: 1; 3
Dietary Supplement: Micronutrients — Zinc 30mg, Magnesium 400mg, Beta-carotene 9 mg, Tocopherol 30mg, vitamin C 200mg y Niacin 100mg.
  Other Names: Intervention II
  Arms: 2; 3
Other: Activities of daily living + placebo — Basic activities of daily living (bathing, dressing, eating, walking) without counseling by a physical therapist and prenatal care.
  Placebo Comparator: Equivalent to placebo (maltodextrin).
  Arms: 4

SUMMARY:
At the moment, most of efforts to prevent non-transmissible chronic diseases at population level have been centered in promoting healthful behaviors like physical activity, consumption of fruits and vegetables, and discouraging from the consumption of tobacco and alcohol in adult population, but the results have been little hopeful. In the last years, manifold studies have indicated the relation between metabolic alterations and of the fetal growth with the development of non-transmissible chronic diseases in adult age. More recently, it has been proposed that maternal factors (endothelial function, oxidative stress and alterations in adipokines) and placental ones (mitochondrial dysfunction) are the precursory mechanisms of fetal metabolic alterations and of the later development of non-transmissible chronic diseases. Also, it has been suggested that possibly supplementation with micronutrients and the physical exercise during the gestation can regulate these maternal and placental factors. For the reasons just mentioned, it is necessary to clarify if these proposed factors are related to fetal metabolic alterations and if the supplementation during the gestation with micronutrients and/or the physical exercise can regulate them, which would be an early and novel alternative to fortify the prevention of non-transmissible chronic diseases in the population.

Purpose

1. To evaluate the effect of associated both the maternal and placental metabolic factors to non-transmissible chronic diseases in newborn.
2. To evaluate the effect of the physical exercise and the complementation with micronutrients during the pregnancy either in the endothelial function, the levels of adipokines, the oxidative stress of the mother and the newborn, as in the placental mitochondrial function and the anthropometry of newborn.

DETAILED DESCRIPTION:
Hypothesis:

1. There is correlation between the metabolic factors, related to non-transmissible chronic diseases, of the mother and those of the newborn one.
2. Supplementation with either micronutrients or physical exercise influence beneficially as much in the endothelial function, oxidative stress, the levels in adipokines of the mother and the newborn one like in the placental mitochondrial function.
3. The simultaneous intervention with micronutrients or physical exercise produces an additional beneficial effect in the metabolic state of the mother and the newborn one.
4. The metabolic alterations when being born are not exclusive of newborn with anthropometric measures located either in the inferior or superior percentiles.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women who have not participated in a structured exercise program, including significant amounts of walking for the past four months are eligible for the trial.
* Live fetus at the routine ultrasound scan and a normal pregnancy.
* Gestational age 16 to 20 weeks
* Written informed consent will be obtained from each woman prior to the inclusion in the study.

Exclusion Criteria:

* History of high blood pressure
* Chronic medical illnesses (cancer, renal, endocrinologic, psychiatric, neurologic, infectious and cardiovascular diseases)
* Persistent bleeding after week 12 of gestation
* Poorly controlled thyroid disease
* Placenta praevia, incompetent cervix, polyhydramnios, oligohydramnios
* History of miscarriage in the last twelve months
* Diseases that could interfere with participation (following recommendations from ACSM 2000, ACOG 2003).

Ages: 16 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 320 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Endothelium-dependent flow mediated dilation | Baseline / week 32-36 of gestation

SECONDARY OUTCOMES:
Biomarkers of endothelial function in blood from umbilical vein and maternal blood | Baseline / 32-36 weeks gestation and delivery
Markers of mitochondrial function | Baseline / 32-36 weeks gestation and delivery
Neonatal and maternal anthropometric indicators | Baseline / 32-36 weeks gestation and delivery
Quality of life SF-12 | Baseline / 32-36 weeks gestation and delivery
Functional capacity (VO2max) | Baseline / 32-36 weeks gestation and delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ana C Plata, MSc, Study Chair — Universidad del Valle, Colombia; Julio Cesar Mateus, MD, MEpi, Study Chair — Fundación FES, División de Salud. Colombia
Locations (1):
- Ana C Plata, MSc, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Derived] Robledo-Colonia AF, Sandoval-Restrepo N, Mosquera-Valderrama YF, Escobar-Hurtado C, Ramirez-Velez R. Aerobic exercise training during pregnancy reduces depressive symptoms in nulliparous women: a randomised trial. J Physiother. 2012;58(1):9-15. doi: 10.1016/S1836-9553(12)70067-X. PMID 22341377
- [Derived] Ramirez-Velez R, Romero M, Echeverri I, Ortega JG, Mosquera M, Salazar B, Giron SL, Saldarriaga W, Aguilar de Plata AC, Mateus JC. A factorial randomized controlled trial to evaluate the effect of micronutrients supplementation and regular aerobic exercise on maternal endothelium-dependent vasodilatation and oxidative stress of the newborn. Trials. 2011 Feb 28;12:60. doi: 10.1186/1745-6215-12-60. PMID 21356082